CLINICAL TRIAL: NCT01107613
Title: Opinion Leaders to Improve Care After COPD or Asthma Emergency Department (ED) Visits.
Brief Title: The Lung Attack Alert Study
Acronym: TLAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00011325
Record Dates: First submitted 2010-04-12; First posted 2010-04-21 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2017-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: opinion leader; COPD; Emergency Department; relapse; follow-up; evidence-based guidelines; Exacerbation of COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emergencies; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Arm (Experimental): Opinion leader educational letter
  Interventions: Behavioral: Opinion leader educational letter
- Control/Standard Care (No Intervention): Regular care

INTERVENTIONS:
Behavioral: Opinion leader educational letter — All patients will receive prednisone X 10 days and antibiotics X 5 days, as well as an opinion leader educational letter sent to the primary care provider outlining the needs of this patient.
  Arms: Intervention Arm

SUMMARY:
This study will enroll patients who present to Emergency Departments (EDs) and have an acute exacerbation of Chronic Obstructive Pulmonary Disease (COPD) or asthma at discharged in one Edmonton ED. Patients will all be provided with evidence-based discharge (prednisone and an antibiotic for COPD and prednisone and inhaled corticosteroids for asthma) and will be randomized to receive enhanced education to the primary care provider or standard care. The investigators' goal is to determine if an opinion leaders' advice will improve chronic care in these patients.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is the 4th leading cause of morbidity and mortality worldwide. COPD is now seen as a disease that is both preventable and treatable. In order to better facilitate treatment for these patients, a number of consensus guidelines have been developed to help physicians in the diagnosis and chronic management of these patients. However, a number of studies have shown that implementation and adherence to the guidelines by physicians, both at the primary care and specialist level, remains poor. Similar argument can be made for asthma: its a common disease, its readily treatable, and guideline compliance is low.

Patients who experience an Acute Exacerbation of COPD (AECOPD) or asthma have an increased risk of serious adverse events, and therefore, must have their management optimized to improve outcomes. These patients most often are evaluated and treated in their local emergency departments (EDs) for the acute episode; however, follow up care is often left to their primary care physician (PCP). The national rate of patient compliance for follow up with their PCP within the first month following an AECOPD is unknown, however, locally, it is only 30%. Similar local statistics are available for asthma From this, it could be inferred that there is a poor rate for any adjustment in chronic management after an AECOPD or acute asthma presentation and therefore an increased risk of future exacerbations.

It is our belief that informing the PCP that their patient experienced an acute COPD or asthma ED presentation, with a form that provides details of the acute management along with an update of the current guideline recommendations, will improve follow up, compliance with current guidelines and the quality of life for patients with COPD or asthma.

ELIGIBILITY:
Inclusion Criteria:

* Appropriately signed and dated informed consent has been obtained;
* ED patients presenting with an acute exacerbation of COPD requiring treatment in the ED;
* Previous physician-diagnosis of COPD (e.g., emphysema, chronic bronchitis or COPD) either previously or within the ED;
* Age > 40 years of age;
* Current or former smokers of more than 10 pack years (number of packs of cigarettes {or pipe and/or cigars) smoked per day X the number of years of smoking);
* FEV1/FVC ratio < 0.7 for age, sex and height (either known or determined within the ED);
* Patients can read and comprehend English language.

Exclusion Criteria:

* Patients presenting for prescription renewal;
* Patients who require hospitalization;
* Patients who do not have a primary care physician or patients for whom a family physician cannot be found;
* Patients who have already been enrolled in the study;
* Patients with a ED physician-diagnosis of primary asthma, pneumonia, HIV/AIDS, immuno-compromise, or life expectance of < 90 days;
* Patients who, in the opinion of the investigator, should be excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Follow-up with primary care provider | 90 days
  The follow-up of the patient by their primary care provider for review of the acute and chronic management of their COPD or asthma and addressing any issues on the Lung Attack Alert, within the first 90 days after discharge from the ED.

SECONDARY OUTCOMES:
Relapse | 90 days
  An unscheduled visit for worsening COPD or asthma symptoms. relapse will be sub-divided into various categories (relapse- no change in management; relapse- change in management; relapse-ED visit change in management and discharged; relapse-ED visit change in management and admission; relapse-death)
Adjusted management | 90 days
  The TLAL letter will identify patients who need review and adjustment of the management of their COPD or asthma (e.g., medication change, smoking cessation strategies, pulmonary rehabilitation, etc). This assessment will document all of the actions taken by the primary care provider after ED discharge.
Length of ED Stay | Up to 24 hours
  The length of stay from the triage to the departure from the ED.
Quality of life | 90 days
  Change in patients' health-related quality of life, within 90 days of discharge from the ED.
Referrals | 90 days
  The numbers of referrals for pulmonary rehabilitation, spirometry, Pulmonary Clinic.
Follow-up with primary care provider | 30 days
  The follow-up of the patient by their primary care provider for review of the acute and chronic management of their COPD and addressing any issues on the Lung Attack Alert, within the first 30 days after discharge from the ED.

CONTACTS AND LOCATIONS:
Overall Officials: Brian H Rowe, MD, MSc, Principal Investigator — University of Alberta; Mohit Bhutani, MD, FRCPC, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta Hospital Emergency Department, Edmonton, Alberta
  - Northeaset Community Health Clinic, Edmonton, Alberta

REFERENCES:
- [Derived] Cross AJ, Thomas D, Liang J, Abramson MJ, George J, Zairina E. Educational interventions for health professionals managing chronic obstructive pulmonary disease in primary care. Cochrane Database Syst Rev. 2022 May 6;5(5):CD012652. doi: 10.1002/14651858.CD012652.pub2. PMID 35514131
- See also: CTS COPD Guidelines — http://www.copdguidelines.ca

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2010-10-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT01107613/Prot_SAP_000.pdf
  • Informed Consent Form (2010-10-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT01107613/ICF_001.pdf